CLINICAL TRIAL: NCT04469400
Title: Study on Lifestyle Intervention for Patients With Impaired Glucose Regulation
Brief Title: Lifestyle Intervention for Patients With Impaired Glucose Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-317
Record Dates: First submitted 2020-06-17; First posted 2020-07-14 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2021-07

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group1 (No Intervention): Researchers conduct health education on patients, including dietary guidance, physical activity guidance, psychological behavior counseling, etc.
- Group2 (Experimental): In addition to education, the subjects will consume 2 composite protein solid drinks per day, in conjunction with the three-meal diet to increase satiety and intake of sufficient nutrients
  Interventions: Dietary Supplement: Low fat diet intensive intervention
- Group3 (Experimental): In addition to education, the subjects will consume 2 nutrition bars daily to replace the staple food of daily lunch and dinner to help reduce carbohydrate intake and intake of sufficient nutrients
  Interventions: Other: Low-Carbon Water Diet Intensive Intervention

INTERVENTIONS:
Dietary Supplement: Low fat diet intensive intervention — education and Compound protein solid beverage
  Arms: Group2
Other: Low-Carbon Water Diet Intensive Intervention — education and Nutrition bar
  Arms: Group3

SUMMARY:
Impaired glucose regulation (IGR) is closely related to overweight/obesity. By studying different dietary patterns (energy-limited diet vs. low-carbohydrate diet) and intensive lifestyle interventions combined with blood glucose monitoring, glucose regulation of overweight/obesity is affected. To improve the blood glucose and related metabolic indexes of patients with impaired (IGR), establish 1-2 clinical intervention programs for impaired glucose regulation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old ② Fasting blood glucose is between 5.6-6.9 mmol/L (100-125mg/dL) or oral glucose tolerance test (OGTT) 2h plasma glucose (2h-PG) is 7.8-11.1 mmol/L (140-200 mg/dL)

  * 24 kg/m2 ≤ BMI ≤ 35 kg/m2

    * Those who are willing to accept assessment and sign informed consent.

Exclusion Criteria:

* Patients diagnosed with diabetes or undergoing diabetes treatment;

  * Receiving drugs or surgery for weight loss at present or in the past 3 months;

    * Receiving corticosteroid or thyroid hormone treatment;

      * Secondary obesity caused by endocrine, genetic, metabolic and central nervous system diseases;

        * Patients with abnormal liver function (alanine aminotransferase or/and aspartate aminotransferase exceeding the upper limit of normal value 3 times); patients with abnormal renal function (serum creatinine exceeding the upper limit of normal value); suffering from kidney disease and other diseases that need to control protein intake;

          * Diseases affecting the digestion and absorption of food (such as chronic diarrhea, constipation, severe gastrointestinal inflammation, active gastrointestinal ulcer, gastrointestinal resection, cholecystitis/cholecystectomy, etc.); ⑦ Suffering from cardiovascular and cerebrovascular diseases, grade 3 hypertension, chronic hepatitis, malignant tumors, anemia, mental illness and memory disorders, epilepsy and other diseases; ⑧ Suffering from infectious diseases such as active tuberculosis and AIDS; ⑨ During pregnancy or lactation; ⑩Patients with physical disabilities and clinicians think it is not suitable to participate in the study (for example, have a serious disease not included in the discharge criteria) or are unwilling to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Fasting blood glucose | ten weeks
Blood glucose 2 hours after meal | ten weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pianhong Zhang, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (8):
- China (8):
  - Cixi People's Hospital, Cixi, Zhejiang
  - Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Jinhua municipal central hospital, Jinhua, Zhejiang
  - Lishui People's Hospital, Lishui, Zhejiang
  - Ningbo Huamei Hospital, University of Chinese Academy of Sciences, Ningbo, Zhejiang
  - Shaoxing People's Hospital, Shaoxing, Zhejiang
  - The first affiliated hospital of Wenzhou medical university, Wenzhou, Zhejiang
  - Yuyao People's Hospital, Yuyao, Zhejiang

IPD SHARING:
Plan to Share IPD: No